CLINICAL TRIAL: NCT01532336
Title: A Multicenter, Randomized Study of the Efficacy and Safety of NVC-422 Ophthalmic Solution for the Treatment of Adenoviral Conjunctivitis
Brief Title: Efficacy and Safety of NVC-422 in the Treatment of Adenoviral Conjunctivitis
Acronym: BAYnovation™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL1104; BAYnovation (Other: NovaBay)
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2014-07

CONDITIONS: Adenoviral Conjunctivitis
Keywords: adenovirus; conjunctivitis; pinkeye
MeSH Terms: conditions — Adenoviridae Infections; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVC-422 Solution, 0.3% (Experimental): Dosed for 10 days
  Interventions: Drug: NVC-422 Solution, 0.3%
- NVC-422 Vehicle Solution (Placebo Comparator): Dosed for 10 days
  Interventions: Drug: NVC-422 Vehicle Solution

INTERVENTIONS:
Drug: NVC-422 Solution, 0.3% — NVC-422 Ophthalmic Solution dropped onto the eye
  Other Names: Auriclosene
  Arms: NVC-422 Solution, 0.3%
Drug: NVC-422 Vehicle Solution — NVC-422 Vehicle Ophthalmic Solution dropped onto the eye
  Arms: NVC-422 Vehicle Solution

SUMMARY:
The purpose of this study is to evaluate the clinical and microbiological efficacy and safety of NVC-422 compared to vehicle for adenoviral conjunctivitis. Adults and children one year of age and older with diagnosis of adenoviral conjunctivitis in at least one eye based upon a positive adenovirus test result using the Aden-Detactor Plus kit (Rapid Pathogen Screening, Inc).

Subjects will be randomly assigned to receive either NVC-422 or Vehicle.

DETAILED DESCRIPTION:
This is a randomized (1:1) double-masked, vehicle-controlled, multi-center, parallel group study with two treatment arms: NVC-422 Ophthalmic Solution 0.33% ("NVC-422") and NVC-422 Vehicle ("Vehicle").

Subjects that meet all inclusion/exclusion criteria will be enrolled into the study, randomized and evaluated at 6 visits:

* Visit 1: Screening, Day 1
* Visit 2: Day 3
* Visit 3: Day 6
* Visit 4: Day 11 End of Treatment (EOT)
* Visit 5: Day 18 Test-of-Cure (TOC)
* Visit 6: Day 42 Follow-up

Subjects were dosed OU for 10 days. Specimens were collected OU at each visit for quantitative PCR adenoviral load and molecular typing.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms of viral conjunctivitis in at least one eye for 3 days or less
* Bulbar conjunctival injection
* Other inclusion criteria per protocol

Exclusion Criteria:

* Presence of subepithelial infiltrates (SEIs) at the Day 1 visit in either eye
* A suspected bacterial, fungal, herpes, Chlamydia or Acanthamoeba co-infection, based on clinical observation
* Other exclusion criteria per protocol

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sustained Clinical Cure | Day 18

CONTACTS AND LOCATIONS:
Overall Officials: David Stroman, Ph.D., Study Director — NovaBay Pharmaceuticals, Inc.
Locations (48):
- United States (24):
  - Glendale, California
  - Los Angeles, California
  - Petaluma, California
  - San Diego, California
  - Fort Myers, Florida
  - Jacksonville Beach, Florida
  - Tampa, Florida
  - Albany, Georgia
  - Kailua, Hawaii
  - Glenview, Illinois
  - Peoria, Illinois
  - Shawnee Mission, Kansas
  - Hazard, Kentucky
  - Winchester, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hicksville, New York
  - Rockville Centre, New York
  - Asheville, North Carolina
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Spartanburg, South Carolina
- Brazil (6):
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Joinville, Santa Catarina
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- India (14):
  - Hyderabad, Andhra Pradesh
  - Ahmedabad, Gujarat
  - Surat, Gujarat
  - Bangalore, Karnataka
  - Thiruvanathapuram, Kerala
  - Mumbai, Maharashtra
  - Daryāganj, New Dehli
  - New Dehli, New Dehli
  - Bikaner, Rajasthan
  - Jaipur, Rajasthan
  - Chennai, Tamil Nadu
  - Salem, Tamil Nadu
  - Visakhapatnam, Vishakhapatnam
  - Kolkata, West Bengal
- Sri Lanka (4):
  - Colombo
  - Kalubowila
  - Negombo
  - Nugegoda